CLINICAL TRIAL: NCT07361991
Title: A Phase Ib/II Study to Evaluate the Safety and Efficacy of IBI363 in Combination With Bevacizumab With or Without Nab-Paclitaxel as Second-Line Therapy in Patients With Advanced Gastric Cancer
Brief Title: IBI363 Plus Bevacizumab With or Without Nab-Paclitaxel for Second-Line Treatment of Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yongxu Jia, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363GC002
Record Dates: First submitted 2025-12-11; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advan'ce'd; Advanced
MeSH Terms: interventions — Bevacizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI363 + Bevacizumab± nab-paclitaxel (Experimental): Phase Ib
  Patients with advanced gastric cancer or gastroesophageal junction adenocarcinoma (GC or GEJC) who have failed prior standard first-line therapy will receive the following treatments:
  IBI363 in combination with bevacizumab± nab-paclitaxel. IBI363 will be administered at a dose of 3 mg/kg Q3W in Cycle 1, followed by a maintenance dose of 1.5 mg/kg Q3W.
  Bevacizumab will be administered at 7.5 mg/kg Q3W. Treatment will continue until disease progression or unacceptable toxicity, whichever occurs first.
  Nab-paclitaxel will be administered at 260 mg/m² Q3W for 4 cycles.
  During the Phase Ib safety lead-in period, patients will be observed for one treatment
  Interventions: Drug: IBI363; Biological: Bevacizumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: IBI363 — IBI363 will be administered as an intravenous infusion at 1.5 mg/kg or 3 mg/kg every 3 weeks (Q3W) in 28-day cycle 1 and 21-day subsequent cycles, in combination with bevacizumab with or without nab-paclitaxel, as second-line therapy for advanced or metastatic gastric or gastroesophageal junction adenocarcinoma.
Biological: Bevacizumab — Bevacizumab 7.5 mg/kg will be administered as an intravenous infusion every 3 weeks (Q3W) in combination with IBI363, with or without nab-paclitaxel, and continued until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined reasons.
Drug: Nab-paclitaxel — Nab-paclitaxel 260 mg/m² will be administered as an intravenous infusion every 3 weeks (Q3W) for up to 4 cycles in combination with IBI363 and bevacizumab in patients in Cohort 2.

SUMMARY:
This study is for patients with advanced or metastatic gastric cancer whose disease has worsened after first-line systemic therapy. IBI363 is an investigational antibody that may help the immune system recognize and attack cancer cells. This trial will evaluate IBI363 in combination with bevacizumab, with or without nab-paclitaxel, as a second-line treatment.

The study has two parts. In the phase Ib part, small groups of patients will receive IBI363 plus bevacizumab with or without nab-paclitaxel to evaluate the safety, side effects, and tolerability of the combination and to determine an appropriate dose for further study. In the phase II part, additional patients will receive the selected regimen to assess the preliminary antitumor activity of IBI363 in combination with bevacizumab ± nab-paclitaxel, including tumor response and other clinical outcomes, as well as to further describe the safety profile. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons defined in the protocol.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent: The patient must voluntarily sign a written informed consent form and be able to comply with the visit schedule and procedures specified in the protocol.
2. Age: 18 to 75 years (inclusive), male or female.
3. Diagnosis and prior therapy:

   * Histologically confirmed advanced gastric or gastroesophageal junction adenocarcinoma (GC or GEJC).
   * Disease progression or intolerance after prior first-line systemic antitumor therapy including immunotherapy.
   * Primary immune resistance: best response during immunotherapy is stable disease (SD) lasting < 12 weeks, or progressive disease (PD).
   * Acquired immune resistance:

1. For patients with PD on immunotherapy: best response during treatment is complete response (CR), partial response (PR), or SD lasting ≥ 12 weeks; 2. For patients who discontinued immunotherapy for reasons other than disease progression and subsequently developed PD: best response during treatment is CR, PR, or SD lasting ≥ 12 weeks, and the interval between last immunotherapy dose and PD is ≤ 6 months.

4. Baseline hematology (within 7 days before first dose of study drug) must meet all of the following:

* Hemoglobin ≥ 90 g/L;
* Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
* Platelet count ≥ 100 × 10⁹/L;
* Eosinophils < 1.5 × upper limit of normal (ULN).

*In this protocol, "baseline" is defined as the last available assessment prior to the first dose of study drug. Within 7 days before blood sampling, patients must not receive blood products (including packed red blood cells, apheresis platelets, cryoprecipitate, etc.), erythropoiesis-stimulating agents, or colony-stimulating factor support.*

5. Baseline serum chemistry (within 7 days before first dose) must meet all of the following:

* Total bilirubin ≤ 1.5 × ULN (patients with total bilirubin > 1.5 × ULN are allowed if conjugated bilirubin ≤ ULN);
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN;
* Serum creatinine ≤ 1.5 × ULN **or** creatinine clearance (CCr) ≥ 45 mL/min, calculated by the Cockcroft-Gault formula using actual body weight;
* Serum albumin ≥ 32 g/L.

  6. Baseline coagulation function (within 7 days before first dose) must meet all of the following:
* International normalized ratio (INR) ≤ 1.5 × ULN (≤ 3 × ULN if on stable anticoagulation therapy);
* Partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (≤ 3 × ULN if on stable anticoagulation therapy).

  7. Baseline urinalysis (within 7 days before first dose)must meet one of the following:
* Urine protein (UPRO) < 2+ by dipstick, **or**
* 24-hour urine protein < 1 g.

  8. At least one measurable lesion as defined by RECIST v1.1 for solid tumors.

  9. ECOG performance status of 0 or 1 (Eastern Cooperative Oncology Group).

  10. Estimated life expectancy ≥ 3 months.

  11. Contraception: Women of childbearing potential and men whose partners are women of childbearing potential must agree to use effective contraception throughout the treatment period and for 6 months after the last dose of study treatment.

Exclusion Criteria

1. Pregnant or breastfeeding women, or women planning to become pregnant before the first dose of study drug, during study treatment, or within 6 months after the last dose.
2. History of active thrombosis, deep venous thrombosis, or pulmonary embolism within 4 weeks before the first dose of study drug, unless adequately treated and considered clinically stable by the investigator.
3. Clinically significant cardiovascular or cerebrovascular disease, including but not limited to:

   * Ventricular arrhythmias or other uncontrolled arrhythmias requiring medical intervention (e.g., anti-arrhythmic therapy);

   * Severe conduction abnormalities (e.g., third-degree atrioventricular block);

   * QT interval corrected by Fridericia (QTcF) ≥ 480 ms;

   * Uncontrolled arterial hypertension despite optimal medical therapy (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);

   * History of myocarditis;

   * Current congestive heart failure requiring treatment;

   * Left ventricular ejection fraction (LVEF) < 50%;

   * New York Heart Association (NYHA) class III or IV heart failure;

   * Acute coronary syndrome (including myocardial infarction or unstable angina), coronary angioplasty, or stent implantation within 6 months prior to the first dose;

   * Cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose;

   * Known active seizure disorders.
4. Interstitial lung disease, pulmonary fibrosis, pneumoconiosis, drug-induced pneumonitis, radiation pneumonitis, or other forms of restrictive lung disease that require corticosteroids or other treatment, or a history of severely impaired pulmonary function.
5. History of atopic constitution, asthma, or atopic dermatitis.
6. Clinically significant pleural effusion, ascites, or pericardial effusion requiring repeated drainage or associated with significant symptoms.
7. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, or immunosuppressive drugs) within 2 years prior to the first dose of study drug. Replacement therapy (e.g., thyroxine, insulin, or physiological replacement doses of corticosteroids for adrenal or pituitary insufficiency) is not considered systemic treatment.
8. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
9. Known hypersensitivity or allergy to study drugs or any of their excipients.
10. History of significant toxicities related to prior immune checkpoint inhibitor therapy that required permanent discontinuation of that treatment.
11. Unresolved toxicities from prior antitumor therapies > Grade 1 (based on NCI CTCAE), with the exception of the following: persistent Grade 2 alopecia, peripheral neuropathy, hypomagnesemia, or other toxicities that are expected to be irreversible but are stable under medical management (e.g., hypothyroidism controlled with replacement therapy, hypertension controlled to <160/100 mmHg with antihypertensive medications).
12. Incomplete recovery from prior surgery, or having undergone any major surgery within 4 weeks before the first dose of study drug.
13. Active, uncontrolled bleeding or known bleeding diathesis.
14. Major gastrointestinal diseases or conditions within 6 months prior to the first dose, including:

    * History of inflammatory bowel disease;

    * ≥ Grade 2 diarrhea occurring within 2 weeks before the first dose;

    * Radiation enteritis.
15. Uncontrolled tumor-related pain or symptomatic hypercalcemia at screening.
16. Known human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) infection, hepatitis C virus (HCV) infection, or active tuberculosis.

    * Patients who are HBsAg-positive and/or hepatitis B core antibody (HBcAb)-positive must have HBV DNA testing. Patients with HBV DNA ≤ 2.5 × 10³ copies/mL or ≤ 500 IU/mL or below the lower limit of detection may be enrolled. HBsAg-positive patients should receive antiviral therapy against HBV throughout study treatment to prevent viral reactivation.
    * Patients who are anti-HBc (+), HBsAg (-), anti-HBs (-), and have undetectable HBV viral load do not require prophylactic antiviral treatment but must be closely monitored for HBV reactivation.
    * Patients with positive HCV serology but negative HCV RNA or HCV RNA below the lower limit of detection may be enrolled.
    * Patients who have completed HCV treatment and have undetectable viral load may be enrolled.
17. Severe or uncontrolled infection, infection requiring systemic intravenous antibiotics, or fever of unknown origin > 38°C within 2 weeks prior to the first dose of study drug.
18. Any other malignancy diagnosed within 5 years before the first dose of study drug, except for adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, carcinoma in situ that has been completely resected, and localized prostate cancer or papillary thyroid carcinoma that has been cured by radical surgery.
19. **Prohibited medications and treatments** (patients must not receive any of the following):

1) IL-2/IL-15-based cytokine therapies. Use of IL-2/IL-15 as a component of adoptive cell therapy or as immune modulation in immunocompromised patients is allowed.

2) Any chemotherapy or small-molecule targeted therapy within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of study drug, without delayed toxicities, with the exception of:

* Use of nitrosourea agents or mitomycin C within 6 weeks prior to the first dose is prohibited.

  3) Any antibody therapy within 4 weeks prior to the first dose of study drug; 4) Participation in any interventional clinical trial involving medical devices or other therapeutic interventions within 2 weeks prior to the first dose; 5) Palliative radiotherapy within 2 weeks prior to the first dose; 6) Live vaccines for prevention of infectious diseases within 4 weeks prior to the first dose; 7) Immunosuppressive or systemic corticosteroid therapy (> 10 mg/day prednisone or equivalent) within 2 weeks prior to the first dose of study drug; 8) Traditional Chinese medicines with definite antitumor effects within 1 week prior to the first dose.

  20. History of significant toxicities related to prior paclitaxel therapy that required permanent discontinuation of that treatment, or any contraindications to study drugs that, in the opinion of the investigator, preclude safe administration of the study treatment.

  21. Any disease, treatment, laboratory abnormality, or history of drug abuse which, in the opinion of the investigator, may compromise patient safety, interfere with informed consent, affect patient compliance, or interfere with the evaluation of the safety of the study drug.

  22. Psychiatric illness, altered mental status, or history of substance abuse that may interfere with the patient's ability to understand the informed consent process and/or complete required study assessments.

  23. Any other condition that, based on known or foreseeable circumstances, in the investigator's judgment would make the patient unable to comply with the protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | From first dose of study treatment until 90 days after the last dose or end of study, whichever occurs first.
  Incidence, severity, and relationship to study treatment of adverse events (AEs), treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs), graded according to NCI CTCAE. Changes from baseline in 12-lead electrocardiogram (ECG), vital signs, physical examination findings, and clinical laboratory test results will also be assessed.
Overall Survival (OS) | 12 months after the last subject participating in
  Overall Survival (OS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1 | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects
Disease Control Rate (DCR) per RECIST v1.1 | 12 months after the last subject participating in
  Disease control rate is defined as the proportion of patients with a best overall response of CR, PR, or stable disease (SD) according to RECIST v1.1 as assessed by investigators.
Time to Response (TTR) | 12 months after the last subject participating in
  Time to response is defined as the time from first dose of study treatment to the date of first documented CR or PR according to RECIST v1.1.
Duration of Response (DoR) | 12 months after the last subject participating in
  Duration of response is defined as the time from the first documented CR or PR to the first documented disease progression or death from any cause, according to RECIST v1.1.
Progression-Free Survival (PFS) | 12 months after the last subject participating in
  Progression-free survival is defined as the time from first dose of study treatment to the first documented disease progression according to RECIST v1.1 or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No